CLINICAL TRIAL: NCT05064410
Title: Screen to Save: NCI Colorectal Cancer Outreach & Screening Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19103; 3P30CA076292-21S3 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Colon Cancer; Cancer prevention
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention and Referral for Fecal Immunochemical Test (FIT) Kit or Colonoscopy (Experimental): The Community Health Educator (CHE) will provide online, phone or in-person colorectal cancer (CRC) early detection, prevention, and screening education to increase knowledge of CRC and the importance of screening. These sessions will be conducted in small in-person sessions, virtually within a group, virtually via a self-paced/self-directed online learning module, or one-on-one via phone. Additionally, the CHE will provide information regarding FIT kit and colonoscopy screening and the screening process for attendees. The CHE and research assistant will be prepared to provide access to screening resources and services through participants' existing coverage. Those participants who do not have a primary care provider will be provided information on obtaining FIT kits through the mechanisms of the Federally Qualified Health Center (FQHC) and/or a colonoscopy through the cancer center on a case by case basis.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — The colorectal cancer (CRC) educational activities will include the use of NCI CRC resources and materials, including a PowerPoint presentation, and CRC educational models and displays. The CRC education will be delivered in Spanish and English, and will consist of pre and post knowledge assessments including screening and behavioral intention questions. The educational intervention will take approximately 45 minutes-1 hour.

SUMMARY:
The purpose of this study is to provide educational materials and information regarding colorectal cancer (CRC), CRC screenings, and United States Preventive Services Task Force's (USPSTF) screening recommendations. USPSTF recommends screening for colorectal cancer starting at age 45 years and continuing until age 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Between 45 and 75 years of age
* Spanish or English speaking
* Able to provide informed consent
* Reside in the Tampa Bay area (namely Hillsborough, Pinellas, Polk or Pasco county)

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge Related to Colorectal Cancer Risk, Prevention, and Screening | Baseline, immediately following intervention, at 3 months and at 6 months
  Pre and post assessment surveys completed by participants will consist of 14 questions assessing knowledge of CRC, risk factors, and screening options and recommendations. Assessments also include 5 questions to determine intentions to change screening/health behaviors, speaking to one's healthcare provider about screening, getting screened, and talking with family/friends about CRC and CRC screening.
  3-month follow up survey consists of 5 sections to determine CRC knowledge, screening behavior since baseline, future screening plans, talking with family and friends about CRC screening, and behavior changes in eating habits and physical activity since partaking in the educational session.
  6-month survey consists of 5 questions about screening since the 3-month follow up survey. Those needing to complete the 6-month follow up survey are those that were screened at the time of the 3-month follow-up but had not received final diagnostic results.

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Gwede, PhD, MPH, RN, FAAN, Principal Investigator — Moffitt Cancer Center; Cathy D Meade, PhD, RN, FAAN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States